CLINICAL TRIAL: NCT04289389
Title: Prevalence and Level of Diagnosis of Dementia in a Population-based Sample in the County of Trøndelag
Status: Active, not recruiting | Type: Observational
Sponsor: Norwegian Centre for Ageing and Health (Other)
Collaborators: Norwegian Health Association (Other); University of Oslo (Other)
Responsible Party: Sponsor
Other Study IDs: 181124
Record Dates: First submitted 2020-02-06; First posted 2020-02-28 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Dementia
Keywords: Prevalence; Epidemiology; Alzheimer's disease
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HUNT4 70+: All inhabitants in Nord-Trøndelag 70 years of age and older were invited.
- HUNT4 Trondheim 70+: All inhabitants of one district in Trondheim 70 years of age and older were invited.

SUMMARY:
To investigate and make valid estimates of the occurrence of dementia and the most common subtypes of dementia in Trøndelag, and transfer these figures to estimates of the occurrence of dementia in Norway as a whole, by age, sex and severity of dementia. Furthermore, the proportion of people without dementia diagnosis among those with dementia will be examined. The investigators will further investigate whether there are differences in dementia prevalence between males and females and educational groups and look at factors associated with a lack of diagnosis.

DETAILED DESCRIPTION:
Introduction There are currently no valid estimates of the occurrence of dementia in Norway. Estimates in use range from 70.000 to 104.000, with the highest estimate being 50 percent greater than the lowest. This makes it difficult to plan today's health services and estimate future needs.

To enable good planning of services to people with dementia, it is important that people with dementia to be evaluated and diagnosed for their illness. An early diagnosis seems to improve prognosis for the course of the disease. The proportion of undiagnosed people with dementia differs in the studies done on this and it is unclear which factors that may explain why many remain undiagnosed for their dementia disease. As a quality measure on the cognitive data being collected in this study we will make population-based Norwegian norms for the Montreal Cognitive Assessment Test (MoCA) test and the Ten-word delayed recall test from CERAD.

The aim of this study is to provide knowledge that is crucial for planning good health and care services for older people with cognitive impairment and dementia. We will make valid estimates for the prevalence of dementia and the most common subtypes of them in Trøndelag and transfer these figures to estimates to Norway as a whole, by age, gender and severity of disease. We will investigate whether there are differences in dementia prevalence between males and females and educational groups. Furthermore, there will be made a survey of the proportion of people without dementia diagnosis among those with dementia, and examine the factors associated with a lack of diagnosis.

Method The data collection was a collaboration with the Health Survey in Nord-Trøndelag when this was carried out for the fourth time (HUNT4) in the period 2017-2019. All persons over the age of 70 living in 23 municipalities in Nord-Trøndelag and a district in Trondheim municipality (Trøndelag) were invited to an assessment at a field stations or by home visits (including institutionalized care), in the study parts called HUNT4 70+ and HUNT4 Trondheim 70+. The participants were offered a survey of cognition and function in everyday life. To get more information on cognitive function an interview with next of kin were made for participants with possible cognitive impairment.

A diagnostic work-up group of scientific and clinical experts (geriatrics, old age psychiatry or neurology) assessed the cases and made the research-based diagnosis. Standard diagnostic criteria according to the DSM-5 was applied for all the dementia diseases. The new estimates from Trøndelag will be used to estimate the occurrence of dementia in Norway as a whole, by age, sex and severity of dementia. Furthermore, the proportion of people without dementia diagnosis among those with dementia will be examined. Information about known dementia diagnosis from dementia assessment in municipality or specialist health service will be obtained by linking to registered data. The investigators will further investigate whether there are differences in dementia prevalence between males and females and educational groups and look at factors associated with a lack of diagnosis. Information from the earlier waves of HUNT (1-4) will be used to get information on health and risk factors for dementia from the study population.

ELIGIBILITY:
Inclusion Criteria:

* Living in the designated area

Exclusion Criteria:

* None

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Persons of 70 years of age or older participated in HUNT4 and accepted cognitive screening in HUNT4 70+.
Sampling Method: Non-Probability Sample
Enrollment: 11675 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dementia criteria in DSM-5 | Each participant is evaluated against dementia criteria in DSM- after participation, based on assessment done in the 20 month long assessment period
  Used to assess prevalence of dementia in the study population

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | Each participant were assessed once during an assessment period of 20 months
  Tests cognitive function in the domain's memory, visuospatial and executive functions, attention, concentration, language and orientation. Scores from 0 - 30 where 30 indicates best function.
CERAD Ten-word test | Each participant is assessed once during an assessment period of 20 months
  Tests immediate and delayed memory. Scores from 0 - 30 in immediate memory and 0-10 in delayed recall, higher scores indicates better function.
Severe Impairment Battery | Participants in institution with known moderate to severe dementia is assessed once during an assessment period of 20 months
  Tests cognitive function in people with moderate to severe dementia. Scores from 0 - 16 where 16 indicates best function.
Hospital Anxiety and Depression Scale | Each participant is assessed once during an assessment period of 20 months.
  Gathers information on anxiety and depression, scores from 0 - 42 where 0 indicates best function
Instrumental Activities in Daily Living Scale | Assessed in proxy interview during interview period of 22 months
  Assess problems with instrumental activities of daily living, scores function in 8 instrumental activities, lower scores indicates better function
Physical Self-Maintenance Scale | 20 months
  Assess problems with personal activities of daily living. Assessed in proxy interview and by health personnel for participants in institutions, scores function in 6 personal activities, lower scores indicates better function
Neuropsychiatric Inventory | 22 months
  Assess neuropsychiatric symptoms, screening questions on each symptom and a score for frequency from 1-4, severity 1-3 and distress 1-5, higher scores indicates more severe symptoms
Clinical Dementia Rating Scale | 22 months
  Assess degree of cognitive decline and function level, scores from 0-3 where higher score indicates more cognitive decline and lower function level

CONTACTS AND LOCATIONS:
Overall Officials: Geir Selbæk, PhD, Principal Investigator — Norwegian National Advisory Unit on Ageing and Health
Locations (1):
- Norwegian National Advisory Unit on Ageing and Health, Tønsberg, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Engedal K, Gjora L, Benth JS, Wagle J, Ronqvist TK, Selbaek G. The Montreal Cognitive Assessment: Normative Data from a Large, Population-Based Sample of Cognitive Healthy Older Adults in Norway-The HUNT Study. J Alzheimers Dis. 2022;86(2):589-599. doi: 10.3233/JAD-215442. PMID 35094994
- [Background] Gjora L, Strand BH, Engedal K, Ernstsen L, Myrstad C, Skjellegrind H, Thingstad P, Selbaek G. Dementia and mild cognitive impairment in older people in Trondelag. Tidsskr Nor Laegeforen. 2023 Jun 26;143(10). doi: 10.4045/tidsskr.22.0815. Print 2023 Jun 27. English, Norwegian. PMID 37376934
- [Background] Wagle J, Selbaek G, Benth JS, Gjora L, Ronqvist TK, Bekkhus-Wetterberg P, Persson K, Engedal K. The CERAD Word List Memory Test: Normative Data Based on a Norwegian Population-Based Sample of Healthy Older Adults 70 Years and Above. The HUNT Study. J Alzheimers Dis. 2023;91(1):321-343. doi: 10.3233/JAD-220672. PMID 36404547
- [Result] GjOra L, Strand BH, Bergh S, Borza T, Braekhus A, Engedal K, Johannessen A, Kvello-Alme M, Krokstad S, Livingston G, Matthews FE, Myrstad C, Skjellegrind H, Thingstad P, Aakhus E, Aam S, Selbaek G. Current and Future Prevalence Estimates of Mild Cognitive Impairment, Dementia, and Its Subtypes in a Population-Based Sample of People 70 Years and Older in Norway: The HUNT Study. J Alzheimers Dis. 2021;79(3):1213-1226. doi: 10.3233/JAD-201275. PMID 33427745
- See also: Website that shows the current and future prevalence of dementia in the different regions and municipalities in Norway — http://demenskartet.no/